CLINICAL TRIAL: NCT05149690
Title: Effectiveness of Monopolar Dielectric Diathermy by Radiofrequency and Supervised Therapeutic Exercise in Pain, Functionality, Mobility of the Spine and Quality of Life of Patients With Non-specific Chronic Low Back Pain.
Brief Title: Monopolar Dielectric Diathermy by Radiofrequency and Therapeutic Exercise in Patients With Chronic Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UALBIO2021/006
Record Dates: First submitted 2021-09-17; First posted 2021-12-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
Keywords: non-specific chronic low back pain; Supervised therapeutic exercise; monopolar dielectric diathermy; randomised single-blind clinical trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monopolar dielectric diathermy and supervised therapeutic exercise (Experimental): The Experimental Group formed by 30 subjects will undergo an application of monopolar electrical diathermy by radiofrequency emission (MDR) using the Physicalm® device developed by the electro-medicine company Biotronic Advance Develops SL, on the lumbar musculature by means of rotary movements and translation, adapting to the muscle fibers of the lumbar area. A pulsed emission of 840 KHz and 30v will be made dynamically during a treatment time of 20 minutes. Once the application of (MDR) is finished, an exercise program supervised by a physiotherapist will be carried out. The exercise program will consist mainly of three types: stability and lumbo-pelvic motor control, strengthening and stretching of the lumbar muscles (Annex XIV), with a duration of 20 minutes. 2 weekly sessions will be held for 4 weeks, distributed as follows: Monday and Wednesday or Tuesday and Thursday, a total of 8 treatment sessions.
  Interventions: Other: Experimental: monopolar dielectric diathermy and supervised therapeutic exercise
- Supervised therapeutic exercise (Active Comparator): The Control Group formed by 30 subjects will be administered a training program consisting of three types of exercises, taking into account: stability and lumbopelvic motor control, strengthening and stretching of the lumbar muscles, exactly the same as the Experimental Group. With a duration of 20 minutes. 2 weekly sessions will be held for 4 weeks, distributed as follows: Monday and Wednesday or Tuesday and Thursday with a total of 8 treatment sessions.
  Interventions: Other: Active Comparator: Supervised therapeutic exercise

INTERVENTIONS:
Other: Experimental: monopolar dielectric diathermy and supervised therapeutic exercise — The Experimental Group formed by 30 subjects will undergo an application of monopolar electrical diathermy by radiofrequency emission (MDR) using the Physicalm® device developed by the electro-medicine company Biotronic Advance Develops SL, on the lumbar musculature by means of rotary movements and translation, adapting to the muscle fibers of the lumbar area. A pulsed emission of 840 KHz and 30v will be made dynamically during a treatment time of 20 minutes. Once the application of (MDR) is finished, an exercise program supervised by a physiotherapist will be carried out. The exercise program will consist mainly of three types: stability and lumbo-pelvic motor control, strengthening and stretching of the lumbar muscles (Annex XIV), with a duration of 20 minutes. 2 weekly sessions will be held for 4 weeks, distributed as follows: Monday and Wednesday or Tuesday and Thursday, a total of 8 treatment sessions.
  Arms: monopolar dielectric diathermy and supervised therapeutic exercise
Other: Active Comparator: Supervised therapeutic exercise — The Control Group formed by 30 subjects will be administered a training program consisting of three types of exercises, taking into account: stability and lumbopelvic motor control, strengthening and stretching of the lumbar muscles, exactly the same as the Experimental Group. With a duration of 20 minutes. 2 weekly sessions will be held for 4 weeks, distributed as follows: Monday and Wednesday or Tuesday and Thursday with a total of 8 treatment sessions.
  Arms: Supervised therapeutic exercise

SUMMARY:
A total of 60 people diagnosed with non-specific chronic low back pain of more than 3 months of evolution and who are not currently undergoing any type of treatment will be recruited, with ages between 30 and 65 years. A random distribution will be made into two treatment groups (diathermy combined with supervised therapeutic exercise versus supervised therapeutic exercise). Participants will receive treatment once a week for a period of four weeks, in the physiotherapy laboratories of the University of Almería, with a follow-up evaluation at three weeks and two months after the start of treatment. At their first visit, participants will be screened for study eligibility according to the study inclusion and exclusion criteria, and will be evaluated by a therapist blinded to the intervention. After this face-to-face evaluation, patients will be randomly assigned to one of the two groups and will receive treatment for low back pain according to their random assignment group by two therapists belonging to the research group and trained in the techniques used.

DETAILED DESCRIPTION:
After randomization, participants will be assigned to the experimental group (8 sessions of monopolar dielectric diathermy by emission of radiofrequency combined with 8 sessions of supervised therapeutic exercise) or to the control group (8 sessions of supervised exercise). The number of participants will be identical between the groups. The randomization sequence will be performed by the principal investigator.

The number of participants for each group will be 30. The results of the random assignment will be sealed in opaque envelopes before being delivered to the participants.

The outcome assessor and study statistician will be blinded throughout the entire process.

A baseline assessment of the primary and secondary outcome measures will be performed before randomization of the participants to the different groups, an immediate post-treatment assessment (1 day after the last intervention) and an assessment two months after the end of the procedure. intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 67 years old.
* Score ≥ 4 points on the Roland Morris Disability Questionnaire.
* Not being receiving physical therapy.

Exclusion Criteria:

(1) patients with sensory and/or coagulation disorders; (2) a history of spinal surgery; (3) heart complications; (4) concurrent severe central or peripheral nervous system disease; (5) epilepsy; (6) needle phobia; (7) serious pathologies that can be the main cause of chronic LBP (for example, presence of lumbar stenosis, spondylolisthesis, tumours, etc.); (8) or patients contraindicated for radiofrequency (diathermy).

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ). | At baseline, at 4 weeks and at 2 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 4 weeks and at 2 months
  It has 10 items associated to activities of daily living, each ítem has a puntuation fron 0 to 5 points.
Change from baseline in pain intensity. Visual analogue scale. | At baseline, at 4 weeks and at 2 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, at 4 weeks and at 2 months
  Is a 17-item questionnaire that measures the fear of movement and (re)injury. Ratings are summed to yield a total score (ranging from 17-68 points) where higher values reflect greater fear of (re)injury.
Change from baseline on Quality of Life. SF-36 Health questionnaire. | At baseline, at 4 weeks and at 2 months
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test. | At baseline, at 4 weeks and at 2 months
  It measures the isometric endurance of trunk flexion muscles.
Change from baseline in lumbar mobility flexion. | At baseline, at 4 weeks and at 2 months
  For the quantification of lumbar flexion an angular inclinometer is used (Fleximeter UM 8320-3 RJ Code Research Institute, Brazil).
Change from baseline in range of motion and lumbar segmental mobility | At baseline, at 4 weeks and at 2 months
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.
Change from baseline of Pittsburgh Sleep Quality Index (PSQI) | At baseline, at 4 weeks and at 2 months
  Is a 10-item questionnaire with a total of 19 questions related to sleep habits in the previous month. The questions are divided into 7 areas, each with a score of between 0 and 3 points.
Change from baseline in Hospital Anxiety and Depression Scale (HADS) | At baseline, at 4 weeks and at 2 months
  assessed the emotional distrees. It consists of two subscales (HADA: anxiety and HADD: depression) with seven items each that score from 0 (normal) to 3 (abnormal)

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

REFERENCES:
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Adamson J, Hunt K, Nazareth I. The influence of socio-demographic characteristics on consultation for back pain--a review of the literature. Fam Pract. 2011 Apr;28(2):163-71. doi: 10.1093/fampra/cmq085. Epub 2010 Oct 25. PMID 20974654
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Haldeman S, Dagenais S. A supermarket approach to the evidence-informed management of chronic low back pain. Spine J. 2008 Jan-Feb;8(1):1-7. doi: 10.1016/j.spinee.2007.10.009. No abstract available. PMID 18164448
- [Background] Lambeek LC, van Tulder MW, Swinkels IC, Koppes LL, Anema JR, van Mechelen W. The trend in total cost of back pain in The Netherlands in the period 2002 to 2007. Spine (Phila Pa 1976). 2011 Jun;36(13):1050-8. doi: 10.1097/BRS.0b013e3181e70488. PMID 21150697
- [Background] Wieser S, Horisberger B, Schmidhauser S, Eisenring C, Brugger U, Ruckstuhl A, Dietrich J, Mannion AF, Elfering A, Tamcan O, Muller U. Cost of low back pain in Switzerland in 2005. Eur J Health Econ. 2011 Oct;12(5):455-67. doi: 10.1007/s10198-010-0258-y. Epub 2010 Jun 5. PMID 20526649
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] van Tulder M, Malmivaara A, Hayden J, Koes B. Statistical significance versus clinical importance: trials on exercise therapy for chronic low back pain as example. Spine (Phila Pa 1976). 2007 Jul 15;32(16):1785-90. doi: 10.1097/BRS.0b013e3180b9ef49. PMID 17632400
- [Background] Kumaran B, Watson T. Thermal build-up, decay and retention responses to local therapeutic application of 448 kHz capacitive resistive monopolar radiofrequency: A prospective randomised crossover study in healthy adults. Int J Hyperthermia. 2015;31(8):883-95. doi: 10.3109/02656736.2015.1092172. Epub 2015 Nov 2. PMID 26524223
- [Background] Úbeda A, Hernández-Bule ML, Trillo MA, Cid MA, Leal J. Cellular response tonon-thermal doses of radiofrequency currents used in electro-thermaltherapy. J Jpn Soc Laser Surg Med. 2006;27(3):187.31.
- [Background] Tashiro Y, Hasegawa S, Yokota Y, Nishiguchi S, Fukutani N, Shirooka H, Tasaka S, Matsushita T, Matsubara K, Nakayama Y, Sonoda T, Tsuboyama T, Aoyama T. Effect of Capacitive and Resistive electric transfer on haemoglobin saturation and tissue temperature. Int J Hyperthermia. 2017 Sep;33(6):696-702. doi: 10.1080/02656736.2017.1289252. Epub 2017 Feb 19. PMID 28139939
- [Background] Kumaran B, Watson T. Radiofrequency-based treatment in therapy- related clinical practice - a narrative review. Part II: chronic conditions. Phys Ther Rev. 2016;20:325-343.
- [Background] Albornoz-Cabello M, Barrios-Quinta CJ, Escobio-Prieto I, Sobrino-Sanchez R, Ibanez-Vera AJ, Espejo-Antunez L. Treatment of Patellofemoral Pain Syndrome with Dielectric Radiofrequency Diathermy: A Preliminary Single-Group Study with Six-Month Follow-Up. Medicina (Kaunas). 2021 Apr 28;57(5):429. doi: 10.3390/medicina57050429. PMID 33925211
- [Background] Ibanez-Vera AJ, Garcia-Romero JC, Alvero-Cruz JR, Lomas-Vega R. Effects of Monopolar Dielectric Radiofrequency Signals on the Symptoms of Fibromyalgia: A Single-Blind Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Apr 3;17(7):2465. doi: 10.3390/ijerph17072465. PMID 32260313